CLINICAL TRIAL: NCT05434806
Title: Estimation of Daily Optimal Efficacy Dose (OED) of Jarlsberg Cheese to Increase the Osteocalcin Level in Healthy Norwegian Elderly Male and Female
Brief Title: Daily Dose Estimation of Jarlsberg Cheese in Healthy Norwegian Elderly Male and Female
Acronym: HV-ID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meddoc (Other)
Collaborators: Tine (Industry)
Responsible Party: Principal Investigator, Prof Stig Larsen, Research Director, Meddoc
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HV-Jarlsberg/ID
Record Dates: First submitted 2022-06-17; First posted 2022-06-28 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Healthy Aging
Keywords: Jarlsberg cheese

STUDY DESIGN:
Intervention Model Description: Between-patients Response Surface Pathway (RSP)
Who Masked: Investigator
Masking Description: Jarlsberg cheese
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post menomausal women (PMW) (Experimental): 40g/day of Jarlsberg cheese will be given three PMW's in the first designlevel. Based on the change in serum osteocalcin level after 4 weeks, the daily Jarlsberg cheese dose for five new PMWs in the second designlevel will be calculated. The results obtained by these five will be used to calculate the dose for seven new PMWs in the third design level.
  Interventions: Dietary Supplement: Jarlsberg cheese
- Men passed the age of 65 years (Experimental): 40g/day of Jarlsberg cheese will be given three men in the first designlevel. Based on the change in serum osteocalcin level after 4 weeks, the daily Jarlsberg cheese dose for five new men in the second designlevel will be calculated. The results obtained by these five will be used to calculate the dose for seven new men in the third design level.
  Interventions: Dietary Supplement: Jarlsberg cheese

INTERVENTIONS:
Dietary Supplement: Jarlsberg cheese — Daly oral intake

SUMMARY:
Aim: To estimate OED of Jarlsberg cheese and the stabilized level of serum Osteocalcin in healthy elderly men and women.

Study population consists of healthy men at least 65 years old and healthy post-menopausal women.

Trial treatment: Daily intake of Jarlsberg cheese within a window of [20 - 100] gram/day and a starting dose of 40 gram/day Design: The study will be performed as an open, two-armed between-patient randomized Response Surface Pathway (RSP) study with three design level and skewed starting dose.

Study procedure: HVs who fulfils the inclusion criteria, do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study one week later. All demographic data, social factors and history of disease will be recorded. The design consists of three design levels and measurement taken at screening, after four weeks daily intake of the decided dose of Jarlsberg cheese. At screening, after four weeks of daily intake of Jarlsberg cheese, a physical examination ,CTCAE and concomitant medication will be performed. Additionally, blood sampling will be taken at screening and after four weeks for measurements of Osteocalcin, PINP, CTX, BALP, vitamin K and common laboratory variables.

Sample size: Fifteen female and 15 male HVs divided on 3 design levels.

DETAILED DESCRIPTION:
Aim: To estimate OED of Jarlsberg cheese and the stabilized level of serum Osteocalcin in healthy elderly men and women.

Study population consists of healthy men at least 65 years old and healthy post-menopausal women.

Trial treatment: Daily intake of Jarlsberg cheese within a window of [20 - 100] gram/day and a starting dose of 40 gram/day

Design: The study will be performed as an open, two-armed between-patient randomized Response Surface Pathway (RSP) study with three design level and skewed starting dose. One arm consists of healthy post-menopausal women and the other of healthy men at least the age of 65years. The two arms will be performed separately in parallel with identical RSP-design.

The aim is to estimate OED based on percent change in the Osteocalcin level from baseline to 4 weeks of daily intake of Jarlsberg cheese. The main outcome variable will be categorized in the following four categories:

1. Low increase in the Osteocalcin level: < 10% the last 4 weeks
2. Moderate Low increase in the Osteocalcin level: [10 - 30% > the last 4 weeks
3. Moderate High increase in the Osteocalcin level: [30 - 50% > the last 4 weeks
4. High increase in the Osteocalcin level: ≥ 50% the last 4 weeks

The design consists of three dose levels. Three HVs in each gender arm will be included in the first design level and all receiving the starting dose of Jarlsberg cheese every day in four weeks. The increase in osteocalcin from baseline to four weeks will be used to calculate the doses for the five HVs of both gender in the second design level. Five patients will be included in the second design level and given the daily doses of Jarlsberg cheese recommended from the results obtained in the first design level. Seven patients will be included on the third design level and given the daily doses of Jarlsberg cheese recommended from the results obtained in the second design level.

The OMT for healthy women in pre-menopausal age was previously estimated at 57-gram Jarlsberg cheese per day. It is unknown if this OED will be larger for men and increase / decrease with age. The initial dose window in this study was set to [20 - 100] gram based on the previous dose-response study in healthy pre-menopausal women.

Based on our prior knowledge, the Osteocalcin follows a quadratic function in Jarlsberg cheese dose. The Osteocalcin seem to increase with increasing dose until a maximum (OED) and reduces for higher intake of the cheese. OED might be below the midpoint of the initial dose window of 60gr/day. To optimize the estimation procedure, the skewed starting dose of 40g/day or 2,5 slices of Jarlsberg cheese will be chosen. This gives an adjusted starting dose window of [20 - 60] gr/day. In case the results from all the three HVs of a given gender in the first design level reports an increase < 10% in the Osteocalcin level, the RSP-procedure recommend a maximum escalation in the daily intake of Jarlsberg cheese for the five new HVs of the given gender in the second design level. The new starting dose-window will then be change with the previously used starting dose as lower boundary. In the present study the adjusted dose-window for the second design level will then be [40 - 70] g/day with the new starting dose of 55g/day. In case the result from the three HVs in the first design level obtained an increase in the osteocalcin level between 10% and 30%, the dose to be used in the second design level will be 45g/day with a dose-window of [40 - 50] g/day. Based on the results obtained at the second design level, the similar procedure will be used to calculate the dose used at the third design level. In case the results obtained at on the design level recommend different doses to be used for the next level, the common RSP procedure will be follows.

Randomization: The three HVs allocated to first design level in each of the two parallel gender arms will all receive 40 g/day in four weeks with osteocalcin measurements after every three weeks. A response-dependant block randomisation procedure will be used based on the results obtained after three weeks. This will be performed for the second design level based on the results obtained in the first design level and at the third design level based on the obtained results in the second.

Main variables: The main response variable will be the change in the total Osteocalcin level after four weeks from baseline. The ratio R0= [Carboxylated / Under carboxylated] Osteocalcin, the bone markers Collagen (CTX-1), Procollagen (PINP) and bone specific ALP (BALB) will be used as secondary variables. Vitamin K1 and K2 including the different fractions MK-7, 8, 9 and 9/4H will be used as supporting variables. The Common Terminology Criteria for Adverse Events version 4.0 (CTCAE) will be used for registration of Adverse Events (AE) and toxicity score.

Study procedure: HVs who fulfils the inclusion criteria, do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study one week later. All demographic data, social factors and history of disease will be recorded at screening. The design consists of three design levels and measurement taken at screening, after four weeks daily intake of the decided dose of Jarlsberg cheese. All the participants will be asked not to change anything in their common intake of food during the study except for replacing other cheese with the received daily dose of Jarlsberg. At screening, after four weeks of daily intake of Jarlsberg cheese, a physical examination including registration of vital signs, CTCAE and concomitant medication will be performed. Additionally, blood sampling will be taken at screening and after four weeks for measurements of Osteocalcin, PINP, CTX, BALP, vitamin K and common laboratory variables.

Sample size: Fifteen female and 15 male HVs divided on 3 design levels [3 + 5 + 7] =15 must be included, perform, and complete the study. In case of a fourth design level, the sample size increases to [3 + 5 + 7 +9] =24. This is the minimum number of patients recommended used in a RSP model.

ELIGIBILITY:
Inclusion Criteria:

* Healthy post-menopausal women and men passed the age of 65years

Exclusion Criteria:

* - Known gastrointestinal disorder
* Abnormal liver or kidney function.
* Diabetes
* Suffering from verified cancer
* Under systemic treatment with corticosteroids or other immunosuppressive drugs the last 3 weeks before start of the trial treatment.
* LDL-cholesterol > 3 mmol/L or Triglyceride > 2 mmol/l
* Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment.
* Lactose intolerance or known milk product allergy
* Not able to understand information.
* Do not want or not able to give written consent to participate in the study.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Serum Osteocalcin level | Week 0
  tOC
Serum Osteocalcin level | Week 4
  tOC

SECONDARY OUTCOMES:
PINP | Week 0
  Procollagen type 1 N-terminal propeptide (PINP)
CTX | Week 0
  C-telopeptide 1 collagen (CTX-1)
PINP | Week 4
  Procollagen type 1 N-terminal propeptide (PINP)
CTX | Week 4
  C-telopeptide 1 collagen (CTX-1)

OTHER OUTCOMES:
cOC | Week 0
  Carboxylated Osteocalcin
cOC | Week 4
  Carboxylated Osteocalcin

CONTACTS AND LOCATIONS:
Overall Officials: Stig E Larsen, PhD, Principal Investigator — Meddoc
Locations (1):
- Skjetten Medical Center, Skjetten, Norway

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and informed consent form are finalized and is available for all the researcher participating in the study.
  The data will be analysed and a clinical study report (CSR) distributed to the members of the research group. Based on this report, a manuscript for publication in an international medical journal will be written
Supporting Information: Study Protocol, ICF
Time Frame: All the data from this study will be available in March 2023 and saved in 5 years